CLINICAL TRIAL: NCT05159960
Title: Optimal Treatment Protocol for Selective Laser Trabeculoplasty - Repeat Trial
Acronym: OSLT-R
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OSLT-R; 277612 (Other: FoU i VGR ID number)
Record Dates: First submitted 2021-11-30; First posted 2021-12-16 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Glaucoma, Open-Angle; Pseudoexfoliation Glaucoma; Ocular Hypertension
Keywords: Selective Laser Trabeculoplasty
MeSH Terms: conditions — Glaucoma, Open-Angle; Exfoliation Syndrome; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The treatment protocol is masked for the patient and for the nurses and optometrists conducting measurement of intraocular pressure during follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 180/low (Experimental): SLT treatment in either half of the trabecular meshwork (180 degrees) consisting of 50+/-5 adjacent laser effects. The energy is adjusted 0,1 mJ below the threshold of formation of micro bubbles.
  Interventions: Procedure: SLT
- 180/high (Experimental): SLT treatment in either half of the trabecular meshwork (180 degrees) consisting of 50+/-5 adjacent laser effects. The energy is adjusted to achieve the formation of micro bubbles at 50-75% of laser effects.
  Interventions: Procedure: SLT
- 360/low (Experimental): SLT treatment in the full circumference of the trabecular meshwork (360 degrees) consisting of 100+/-10 adjacent laser effects. The energy is adjusted 0,1 mJ below the threshold of formation of micro bubbles.
  Interventions: Procedure: SLT
- 360/high (Experimental): SLT treatment in the full circumference of the trabecular meshwork (360 degrees) consisting of 100+/-10 adjacent laser effects. The energy is adjusted to achieve the formation of micro bubbles at 50-75% of laser effects.
  Interventions: Procedure: SLT

INTERVENTIONS:
Procedure: SLT — A drop of Pilocarpine 4% is administered to the eye 20 minutes before SLT. Immediately before SLT a drop of Tetracaine hydrochloride 1% is administered. Selective laser trabeculoplasty is conducted through a Latina lens, in a fashion determined by randomization to a study arm (see description).

SUMMARY:
Glaucoma is a common eye disease that can lead to blindness. The only known way to reduce the rate of disease progression is by reducing the pressure in the eye (the intraocular pressure, IOP). Selective laser trabeculoplasty (SLT) is an ophthalmic laser intervention with the purpose of reducing the IOP.

SLT can be performed in different ways, with four of the treatment protocols being evaluated in the Optimal SLT (OSLT) trial.

SLT is a repeatable procedure, but scientific evidence is scarce regarding more than one repetition. In this trial, patients included in the OSLT trial will be invited to the extended trial (OSLT-R), for further follow-up and re-treatment with SLT, if needed.

DETAILED DESCRIPTION:
Subjects already included in the OSLT trial (NCT03798223) will be invited to the extended trial (OSLT-R) at the time of SLT re-treatment or when OSLT follow up is scheduled to terminate. Patients are re-treated as needed, according to the randomized group assignment performed in the OSLT inclusion process.

The OSLT-R trial is aiming to elucidate:

* If the SLT efficacy, in terms of relative IOP reduction (percent of baseline IOP), changes with additional SLT iterations.
* If the longevity of IOP reduction after SLT changes with additional SLT iterations.
* If repeated SLT is associated with a change in postoperative discomfort or adverse events.

All of the above will be analyzed within each of the four treatment groups (SLT protocols) in the trial. Further, analysis will also be conducted regarding differences between the treatment groups regarding the above.

Further, analysis will be performed regarding SLT efficacy depending of the total number of SLT:s an eye has received, including those performed before entering the OSLT and OSLT-R trials.

ELIGIBILITY:
Inclusion Criteria:

* Included in the OSLT trial
* Followed up without the need for other treatment escalation than repeat SLT

Exclusion Criteria:

* Unable to participate in follow up due to health conditions, strength or physical location.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Relative IOP reduction for each SLT iteration | 1-6 months after each SLT, as described above
  Relative IOP reduction for each SLT iteration is calculated as the percentage IOP reduction from baseline (the mean of 3 pre-SLT measurements) to result IOP (the mean of the IOP at follow-up 1, 3 and 6 months after SLT).

SECONDARY OUTCOMES:
Survival (for each SLT iteration) | From randomization to failure (IOP lowering intervention, except repeat SLT) or censoring (death, patients choice), assessed until the last of: 1. 3 years after randomization; 2. 31 Dec 2024 or; 3. Six months after the last SLT during that timespan.
  Kaplan-Meier survival analysis will be conducted, measuring the proportion of eyes that stay in the study groups but do not receive any further IOP-lowering intervention, including repeat SLT.
Survival (repeat SLT allowed) | From each SLT iteration to failure (IOP lowering intervention incl. repeat SLT) or censoring (death, patients choice), assessed until the last of: 1. 3 years after randomization; 2. 31 Dec 2024 or; 3. Six months after the last SLT during that timespan.
  Kaplan-Meier survival analysis will be conducted, measuring the proportion of eyes that stay in the study groups but do not receive any further IOP-lowering intervention, except repeat SLT.
Achievement of 20% reduction in IOP | From randomization until the last of: 1. 3 years after randomization; 2. 31 Dec 2024 or; 3. Six months after the last SLT during that timespan.
  The proportion of eyes achieving and maintaining an IOP reduction of at least 20% compared to baseline.
Absolute IOP reduction for each SLT iteration | 1-6 months after each SLT, as described above
  Absolute IOP reduction for each SLT iteration is calculated as the IOP reduction, in mmHg, from baseline (the mean of 3 pre-SLT measurements) to result IOP (the mean of the IOP at follow-up 1, 3 and 6 months after SLT).
Pain perioperatively: on a scale | Immediately after treatment
  The patient will grade perioperative pain on an arbitrary scale between 0 (no pain) and 4 (maximum pain) on a written protocol.
Pain postoperatively: on a scale | During the first month
  The patient will grade post-operative pain on an arbitrary scale between 0 (no pain) and 4 (maximum pain) on a written protocol, also stating the duration of pain.
Light sensitivity postoperatively: on a scale | During the first month
  The patient will grade post-operative sensitivity to light on an arbitrary scale between 0 (no difference) and 4 (very intense sensitivity to light) on a written protocol, also stating the duration of light sensitivity.
Impairment of vision postoperatively: on a scale | During the first month
  The patient will grade post-operative impairment of vision on an arbitrary scale between 0 (no difference) and 4 (cannot see ones own hand) on a written protocol, also stating the duration of vision impairment.
Redness postoperatively: on a scale | During the first month
  The patient will grade post-operative redness of the eye on an arbitrary scale between 0 (no difference) and 4 (very intense redness) on a written protocol, also stating the duration of redness.
Adverse events | From randomization until the last of: 1. 3 years after randomization; 2. 31 Dec 2024 or; 3. Six months after the last SLT during that timespan. However, generally adverse events are anticipated to emerge in the first post-operative days or weeks.
  The type and frequency of adverse events will be recorded and analyzed in each of the study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Dahlgren, MD, Principal Investigator — Vastra Gotaland Region; Marcelo Ayala, MD, PhD, Study Chair — Vastra Gotaland Region
Locations (2):
- Sweden (2):
  - Department of Ophthalmology, Skaraborg Hospital, Skövde, Västra Götaland County
  - Department of Ophthalmology, NU Hospital Group, Uddevalla, Västra Götaland County

IPD SHARING:
Plan to Share IPD: No